CLINICAL TRIAL: NCT03948386
Title: A Randomized, Controlled, Double-Blind Trial of 3 Local Anesthetics for Spinal Anesthesia in Primary Total Hip Arthroplasty to Compare the Percentage of Patients in Each Group With Early Ambulation
Brief Title: 3 Local Anesthetics for Spinal Anesthesia in Primary Total Hip Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19D.299
Record Dates: First submitted 2019-05-08; First posted 2019-05-13 (Actual); Results first posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-04

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: Patients who agree to participate will then be randomized by a computer-generated sequence to one of the three study groups.
  Dosing will be as follows: isobaric bupivacaine 12.5 mg (2.5 cc of 0.5%) for ≤ 74" height and 15 mg (3 cc) for > 74" height; hyperbaric bupivacaine 10.25 mg (1.5 cc 0.75%) for ≤ 74" height and 13.125 mg (1.75 cc) for > 74" height; and isobaric mepivacaine 52.5 mg (3.5 cc of 1.5%) for ≤ 74" height and 60 mg (4 cc) for > 74" height.
Who Masked: Participant, Outcomes Assessor
Masking Description: The anesthesiologist and certified registered nurse anesthetist or resident performing the spinal will be aware of group allocation and will perform spinal anesthesia according to standard operating procedures with the assigned local anesthetic.
  Patients will remain blinded and surgeons and those performing postoperative assessments will remain blinded as well.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- isobaric bupivacaine (Active Comparator): Isobaric bupivacaine 12.5 mg (2.5 cc of 0.5%) for ≤ 74" height and 15 mg (3 cc) for > 74" height
  Interventions: Drug: isobaric bupivacaine
- hyperbaric bupivacaine (Active Comparator): hyperbaric bupivacaine 10.25 mg (1.5 cc 0.75%) for ≤ 74" height and 13.125 mg (1.75 cc) for > 74" height
  Interventions: Drug: hyperbaric bupivacaine
- isobaric mepivacaine (Active Comparator): isobaric mepivacaine 52.5 mg (3.5 cc of 1.5%) for ≤ 74" height and 60 mg (4 cc) for > 74" height
  Interventions: Drug: isobaric mepivacaine

INTERVENTIONS:
Drug: isobaric bupivacaine — The anesthesiologist and CRNA or resident performing the spinal will perform spinal anesthesia according to standard operating procedures with the randomly assigned local anesthetic.
  Arms: isobaric bupivacaine
Drug: hyperbaric bupivacaine — TThe anesthesiologist and CRNA or resident performing the spinal will perform spinal anesthesia according to standard operating procedures with the randomly assigned local anesthetic.
  Arms: hyperbaric bupivacaine
Drug: isobaric mepivacaine — The anesthesiologist and CRNA or resident performing the spinal will perform spinal anesthesia according to standard operating procedures with the randomly assigned local anesthetic.
  Arms: isobaric mepivacaine

SUMMARY:
Spinal anesthesia is commonly utilized for hip replacement surgery. Different medications used for spinal anesthesia work for different lengths of time. This study will compare three different spinal anesthesia medications in patients having hip replacement surgery to see if patients are able to get out of bed and walk earlier after surgery with one medication versus the others.

DETAILED DESCRIPTION:
Total hip replacement is often performed under spinal anesthesia, which is the standard at Thomas Jefferson University Hospital (TJUH) and Rothman Orthopedic Specialty Hospital (ROSH) for patients without contraindications. Spinal anesthesia involves injecting a numbing medicine (local anesthetic) into the cerebrospinal fluid that bathes the spinal cord through a space between two bones in the back. This causes temporary numbness of the legs and hips and allows surgery to take place without patients feeling pain during surgery. Different local anesthetics can be used for spinal anesthesia and each works for a different duration of time. Another factor that affects how spinal anesthesia medications work is the baricity of the medication, which refers to how dense it is compared to cerebrospinal fluid (CSF). Medications that are less dense than CSF are hypobaric, those with same density are isobaric, and those with greater density are hyperbaric. For clinical purposes, this really only comes into play when positioning the patient immediately after spinal placement as patient position has different effects on the dermatomal level attained depending on baricity of the local anesthetic. Bupivacaine is a long-acting local anesthetic that has been used for several decades for total hip replacement. It is available in both hyperbaric form (with dextrose added) and isobaric form (with no dextrose added). Mepivacaine is another local anesthetic that has a shorter duration of action and is also used for spinal anesthesia in total hip replacement at many centers. All three drugs are used routinely at different centers in the United States. Despite the differences in duration that have been described from pharmacokinetic studies, a randomized, controlled study comparing the three drugs in terms of important outcomes, such as the ability to walk after surgery, has not been published yet. Therefore, the investigators want to compare the three local anesthetics in a randomized, controlled fashion to see if more patients are able to walk sooner after receiving mepivacaine spinal anesthesia than either form of bupivacaine spinal anesthesia.

Patients who are eligible will be called the night prior to surgery and the study will be explained over the phone. Patients who express interest will be recruited on the day of their scheduled surgery in the short-procedure unit. Patients will be given consent forms and time to read them and ask questions.

Preoperative Management All patients without contraindications or allergies will receive oral gabapentin and acetaminophen in the short procedure unit prior to surgery per routine practice.

Intraoperative Management The targeted spinal dermatome level to achieve will be T10 (umbilicus). For isobaric drugs, patients will sit after spinal placement for 3-5 minutes to achieve this level. For hyperbaric bupivacaine, patients will be immediately placed supine and in Trendelenberg position for 3-5 minutes to achieve adequate level and confirmed with sensory pinprick testing, which will be performed every 2 minutes beginning at spinal placement time. After spinal is placed, sedation will be titrated at the discretion of the anesthesia team to achieve the American Society of Anesthesiology's definition of moderate sedation (purposeful response to verbal or tactile stimulation, spontaneous ventilation, and no airway intervention needed) using propofol. All patients will receive tranexamic acid unless contraindicated (10 mg/kg bolus), as well as multimodal analgesia with a non-steroidal anti-inflammatory drug (NSAID) and dexamethasone 4 mg IV per routine practice.

Postoperative Management

Sensory and motor assessments will take place every 30 minutes from PACU arrival time until motor strength is 5/5 in both lower extremities in hip flexion, knee extension, and toe dorsiflexion or the patient's motor function returns to baseline. The time of return of motor function will be documented. Physical therapists will visit the patient between 3 and 3.5 hours after spinal placement to assess for ability to ambulate and perform Tinnetti test, which assesses ambulation and gait and gives a score of 0 through 28 (see attached). Urinary retention will be assessed through asking the following on postoperative day 1:

1. At what time did the participant first urinate?
2. Did participant require a Foley catheter or straight catheter to drain urine from his or her bladder?

These questions will be asked along with the following about TNS (transient neurological symptoms):

1. Does the participant have any pain in his or her lower back that goes into his or her buttocks and/or down his or her thigh that was not there before surgery?
2. If yes, how would the participant rate that specific pain from 0 (no pain) to 10 (worst pain imaginable).
3. How would the participant rate his/her overall pain (0 to 10 scale)?
4. How satisfied is the participant with his/her anesthesia experience (0 to 10 scale where 0 is very dissatisfied and 10 is very satisfied)?

TNS will be defined as the new onset (within 24 hours of surgery) of back pain that radiates into the buttocks, thighs, hips, or distally. Localized back pain will not be included.

Urinary retention will be defined by inability to urinate within 8 hours, a report of distended or painful bladder occurring on postoperative days 0 or 1, either by patient report or on assessment by nursing, or the use of a Foley catheter or straight catheter.

Post-discharge phone calls

The following will be asked to patients via phone calls after discharge at 24 and 48 hours after surgery if not still in the hospital (will be asked in-person otherwise):

1. Does the participant have any back pain that was not present before surgery that goes into his/her buttocks, thighs, hips, or lower leg?
2. If yes, how would the participant rate that specific pain from 0 (no pain) to 10 (worst pain imaginable).
3. How would the participant rate his/her overall pain (0 to 10 scale)?
4. How satisfied is the participant with his/her anesthesia experience (0 to 10 scale where 0 is very dissatisfied and 10 is very satisfied)?

Post-discharge data collection Readmissions within 90 days will be recorded for all patients including the reason for readmission.

General Operating Procedures Patients who agree to participate will then be randomized by a computer-generated sequence to one of the three study groups. The anesthesiologist and certified registered nurse anesthetist or resident performing the spinal will be aware of group allocation and will perform spinal anesthesia according to standard operating procedures with the assigned local anesthetic. Intraoperative sedation will be with propofol or dexmedetomidine, at the discretion of the anesthesia team. Patients will remain blinded and surgeons and those performing postoperative assessments will remain blinded as well. As all study drugs are standard spinal anesthesia drugs and readily available, the anesthesia team caring for the patient will be informed of group allocation and the appropriate drug will be selected. These doses of hyperbaric and isobaric bupivacaine are considered "low dose" and are lower than those routinely used at TJUH and ROSH. However, existing evidence shows that low-dose bupivacaine for spinal anesthesia provides adequate anesthesia time for a total joint replacement. Dosing will be as follows: isobaric bupivacaine 12.5 mg (2.5 cc of 0.5%) for < 74" height and 15 mg (3 cc) for > or = 74" height; hyperbaric bupivacaine 10.25 mg (1.5 cc 0.75%) for < 74" height and 13.125 mg (1.75 cc) for > or = 74" height; and isobaric mepivacaine 52.5 mg (3.5 cc of 1.5%) for < 74" height and 60 mg (4 cc) for > or = 74" height. Patients with BMI of 35 or greater will also be given the higher dose of each of the 3 medications listed above.

Intraoperative variables that will be measured include: hypotension (defined as a decrease in baseline blood pressure of 20% or greater), surgeon rating of intraoperative muscle tension (0, 1, 2, or 3 where 0 is the most relaxed and 3 is the tightest), and conversion to general anesthesia.

Postoperative variables that will be measured include: ambulation at 3-3.5 hours (primary endpoint), time to ambulation, attempts needed to ambulate, episodes of orthostatic hypotension while trying to ambulate, urinary retention, opioid consumption, pain, incidence of transient neurological symptoms up to 48 hours postoperatively, discharge readiness, and length of stay.

Post-discharge phone calls

The following will be asked to patients via phone calls after discharge on postoperative days 1 and 2 after surgery if not still in the hospital (will be asked in-person otherwise):

1. Does the participant have any pain in his/her lower back that goes into his/her buttocks and/or down his/her thigh that was not there before surgery?
2. If yes, how would the participant rate that specific pain from 0 (no pain) to 10 (worst pain imaginable).
3. How would the participant rate his/her overall pain (0 to 10 scale)?
4. How satisfied is the participant with his/her anesthesia experience (0 to 10 scale where 0 is very dissatisfied and 10 is very satisfied)?

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective primary hip replacement surgery
* American Society of Anesthesiologists physical status 1-3

Exclusion Criteria:

* hip fracture
* contraindication to spinal anesthesia (refusal, coagulopathy or recent use of anticoagulant medication that prevents spinal anesthesia, local or systemic infection)
* any other reason deemed significant by attending anesthesiologist
* any patient requiring a wheelchair for ambulation or who cannot walk 25 feet with or without an assist device at time of surgery
* presence of neuropathy in posterior thighs or buttocks
* use of greater than the equivalent of morphine 25 mg IV (oxycodone 30 mg PO) daily
* any patient deemed a poor candidate for spinal anesthesia as determined by the attending anesthesiologist

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Schwenk, MD, Principal Investigator — Thomas Jefferson University
Locations (2):
- United States (2):
  - Rothman Orthopedic Specialty Hospital, Bensalem, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Basques BA, Toy JO, Bohl DD, Golinvaux NS, Grauer JN. General compared with spinal anesthesia for total hip arthroplasty. J Bone Joint Surg Am. 2015 Mar 18;97(6):455-61. doi: 10.2106/JBJS.N.00662. PMID 25788301
- [Background] Kamel HK, Iqbal MA, Mogallapu R, Maas D, Hoffmann RG. Time to ambulation after hip fracture surgery: relation to hospitalization outcomes. J Gerontol A Biol Sci Med Sci. 2003 Nov;58(11):1042-5. doi: 10.1093/gerona/58.11.m1042. PMID 14630887
- [Background] Oldmeadow LB, Edwards ER, Kimmel LA, Kipen E, Robertson VJ, Bailey MJ. No rest for the wounded: early ambulation after hip surgery accelerates recovery. ANZ J Surg. 2006 Jul;76(7):607-11. doi: 10.1111/j.1445-2197.2006.03786.x. PMID 16813627
- [Background] Mahan MC, Jildeh TR, Tenbrunsel TN, Davis JJ. Mepivacaine Spinal Anesthesia Facilitates Rapid Recovery in Total Knee Arthroplasty Compared to Bupivacaine. J Arthroplasty. 2018 Jun;33(6):1699-1704. doi: 10.1016/j.arth.2018.01.009. Epub 2018 Jan 16. PMID 29429882
- [Background] Uppal V, Retter S, Shanthanna H, Prabhakar C, McKeen DM. Hyperbaric Versus Isobaric Bupivacaine for Spinal Anesthesia: Systematic Review and Meta-analysis for Adult Patients Undergoing Noncesarean Delivery Surgery. Anesth Analg. 2017 Nov;125(5):1627-1637. doi: 10.1213/ANE.0000000000002254. PMID 28708665
- [Background] Pawlowski J, Orr K, Kim KM, Pappas AL, Sukhani R, Jellish WS. Anesthetic and recovery profiles of lidocaine versus mepivacaine for spinal anesthesia in patients undergoing outpatient orthopedic arthroscopic procedures. J Clin Anesth. 2012 Mar;24(2):109-15. doi: 10.1016/j.jclinane.2011.06.014. Epub 2012 Feb 17. PMID 22342508
- [Background] Pawlowski J, Sukhani R, Pappas AL, Kim KM, Lurie J, Gunnerson H, Corsino A, Frey K, Tonino P. The anesthetic and recovery profile of two doses (60 and 80 mg) of plain mepivacaine for ambulatory spinal anesthesia. Anesth Analg. 2000 Sep;91(3):580-4. doi: 10.1097/00000539-200009000-00015. PMID 10960380
- [Background] Liguori GA, Zayas VM, Chisholm MF. Transient neurologic symptoms after spinal anesthesia with mepivacaine and lidocaine. Anesthesiology. 1998 Mar;88(3):619-23. doi: 10.1097/00000542-199803000-00010. PMID 9523803
- [Background] YaDeau JT, Liguori GA, Zayas VM. The incidence of transient neurologic symptoms after spinal anesthesia with mepivacaine. Anesth Analg. 2005 Sep;101(3):661-665. doi: 10.1213/01.ane.0000167636.94707.d3. PMID 16115971

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient assigned to isobaric bupivacaine received hyperbaric bupivacaine (miscommunication); two patients assigned to mepivacaine did not receive correct drug from miscommunication; and one patient assigned to hyperbaric bupivacaine was given the wrong drug from miscommunication. One patient assignment information is unclear.
Groups:
- Hyperbaric Bupivacaine: hyperbaric bupivacaine 10.25 mg (1.5 cc 0.75%) for ≤ 74" height and 13.125 mg (1.75 cc) for > 74" height
  hyperbaric bupivacaine: The anesthesiologist and CRNA or resident performing the spinal will perform spinal anesthesia according to standard operating procedures with the randomly assigned local anesthetic.
Period: Overall Study
Arm/Group | Isobaric Bupivacaine | Hyperbaric Bupivacaine | Isobaric Mepivacaine
Started | 52 | 54 | 53
Completed | 51 | 53 | 50
Not Completed | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Baseline data unavailable for the 5 patients out of the 159 who were not included in analyses so 154 were analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Isobaric Bupivacaine | Hyperbaric Bupivacaine | Isobaric Mepivacaine | Total
Number analyzed (Participants) | 51 | 53 | 50 | 154
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 19 | 21 | 64
  >=65 years | 27 | 34 | 29 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (9) | 67 (8) | 67 (8) | 67 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 22 | 78
  Male | 23 | 25 | 28 | 76
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 51 | 53 | 50 | 154

OUTCOME MEASURES:

1. Primary Outcome: Percentage Ambulating Early After Spinal Anesthesia
Description: Is there a difference between isobaric mepivacaine, hyperbaric bupivacaine, and isobaric bupivacaine when used for spinal anesthesia in primary total hip replacement in percentage of patients that can ambulate within 3.5 hours after spinal anesthesia?
Time Frame: 3.5 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Isobaric Bupivacaine | Hyperbaric Bupivacaine | Isobaric Mepivacaine
Number analyzed (Participants) | 51 | 53 | 50
Participants | 9 | 20 | 35

2. Secondary Outcome: Return of Motor Function of the Thigh and Lower Leg
Description: time to return of motor function of the thigh and lower leg
Time Frame: Postoperative day 0 (day of surgery)
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Isobaric Bupivacaine | Hyperbaric Bupivacaine | Isobaric Mepivacaine
Number analyzed (Participants) | 51 | 53 | 50
minutes | 148 [120 to 205] | 123 [88 to 188] | 109 [74 to 156]

3. Secondary Outcome: Number of Patients With Dizziness Events
Description: number of patients with dizziness when transitioning from lying down to sitting or standing
Time Frame: Postoperative day 2
Population: 2 patients with missing data
Measure: Count of Participants; unit: Participants
Arm/Group | Isobaric Bupivacaine | Hyperbaric Bupivacaine | Isobaric Mepivacaine
Number analyzed (Participants) | 51 | 52 | 49
Participants | 11 | 7 | 9

4. Secondary Outcome: Number of Patients With Urinary Retention Events
Description: number of patients with inability to urinate within 8 hours of surgery OR a report of distended or painful bladder occurring on postoperative day 0 or 1, either by patient report or on palpation by nursing
Time Frame: postoperative day 1
Population: 3 patients with missing data
Measure: Count of Participants; unit: Participants
Arm/Group | Isobaric Bupivacaine | Hyperbaric Bupivacaine | Isobaric Mepivacaine
Number analyzed (Participants) | 49 | 52 | 50
Participants | 6 | 8 | 5

5. Secondary Outcome: Number of Patients With Transient Neurological Symptoms (TNS)
Description: Number of patients with TNS events occurring. Transient neurological symptoms were defined as new onset of back, buttock, or thigh pain occurring after spinal anesthesia.
Time Frame: Postoperative days 0-2
Population: Number of patients experiencing TNS at any time.
Measure: Count of Participants; unit: Participants
Arm/Group | Isobaric Bupivacaine | Hyperbaric Bupivacaine | Isobaric Mepivacaine
Number analyzed (Participants) | 51 | 53 | 50
Participants | 2 | 6 | 5

6. Secondary Outcome: Hospital Stay
Description: length of hospital stay
Time Frame: hospital stay (0-3 days)
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Isobaric Bupivacaine | Hyperbaric Bupivacaine | Isobaric Mepivacaine
Number analyzed (Participants) | 51 | 53 | 50
hours | 26 [21 to 28] | 26 [23 to 29] | 22 [9 to 26]

ADVERSE EVENTS:
Time Frame: 3 days
Arm/Group | Isobaric Bupivacaine | Hyperbaric Bupivacaine | Isobaric Mepivacaine
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/53 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/53 | 0/50
Other Adverse Events (participants affected / at risk) | 2/51 | 6/53 | 5/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Isobaric Bupivacaine (N=51) | Hyperbaric Bupivacaine (N=53) | Isobaric Mepivacaine (N=50)
Transient neurologic symptoms (Nervous system disorders) | 2 | 6 | 5 — Response to the question ""Do you have any back pain that you didn't have before surgery that goes into your buttocks, thighs, hips, or lower legs?"

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT03948386/Prot_SAP_000.pdf